CLINICAL TRIAL: NCT01548651
Title: Effect of Saxagliptin Treatment on Myocardial Fat Content, Left Ventricular Function, and Monocyte Inflammation in Patients With Impaired Glucose Tolerance
Brief Title: Effect of Saxagliptin Treatment on Myocardial Fat Content, and Monocyte Inflammation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty with enrollment of subjects
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mandeep Bajaj, Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-29171
Record Dates: First submitted 2012-02-06; First posted 2012-03-08 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo 5 mg orally daily for 6 months
  Interventions: Drug: Placebo
- Saxagliptin (Experimental): Saxagliptin 5 mg orally daily for 6 months
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — Subjects will be randomized to receive either Saxagliptin 5mg daily orally or placebo for 6 months. All subjects will receive baseline measurements of fasting plasma glucose, free fatty acids, plasma adipocytokines, plasma levels of inflammatory markers and C Reactive Protein (CRP), Intracellular Adhesion Molecule (ICAM), vascular cell adhesion molecule (VCAM), plasma lipids, and glucose tolerance (75 gram oral glucose tolerance test) as well as measurement of liver and myocardial fat content and left ventricular systolic and diastolic function with magnetic resonance imaging/spectroscopy. All subjects will also undergo measurements of monocyte inflammatory proteins at baseline. All subjects will undergo repeat measurements of fasting plasma glucose, Free Fatty Acids, inflammatory markers and adipocytokines, oral glucose tolerance test, monocyte inflammation, as well as hepatic/myocardial fat content determination and left ventricular function at the end of the 6 months.
  Other Names: Onglyza
  Arms: Saxagliptin
Drug: Placebo — Subjects will be randomized to receive either Saxagliptin 5mg daily orally or placebo for 6 months. Prior to randomization, all subjects will receive baseline measurements of fasting plasma glucose, free fatty acids, plasma adipocytokines, plasma levels of inflammatory markers and CRP, ICAM, VCAM, plasma lipids, and glucose tolerance (75 gram oral glucose tolerance test) as well as measurement of liver and myocardial fat content and left ventricular systolic and diastolic function with magnetic resonance imaging/spectroscopy. All subjects will also undergo measurements of monocyte inflammatory proteins at baseline. All subjects will undergo repeat measurements of fasting plasma glucose, Free Fatty Acids, inflammatory markers and adipocytokines, oral glucose tolerance test, monocyte inflammation, as well as hepatic/myocardial fat content determination and left ventricular function at the end of the 6 month treatment period.
  Arms: Placebo

SUMMARY:
The purpose of the study is to examine the effect of saxagliptin, an anti-diabetes medication, on hepatic and myocardial fat content and monocyte inflammation in patients with Impaired Glucose Tolerance (IGT).

DETAILED DESCRIPTION:
Obese, insulin resistant individuals have an excess of fat in the liver which is not attributable to alcohol or other known causes of liver disease, a condition defined as nonalcoholic fatty liver disease (NAFLD). The fatty liver is insulin resistant. Individuals with a fatty liver are more likely to have excess intra-abdominal fat as well as a reduction in circulating plasma adiponectin levels. A new class of antidiabetes medications known as dipeptidyl peptidase 4 (DPP-4) inhibitors (sitagliptin, saxagliptin) which enhance the circulating half life of Glucagon-like peptide-1 (GLP-1), an incretin hormone that enhances insulin secretion/ lowers glucose levels, have been approved to treat type 2 diabetes. More recently, it has been shown that these dipeptidyl peptidase 4 inhibitors can also decrease liver fat and inflammation in animal models of obesity by increasing circulating levels of GLP-1. It has been shown that GLP-1 enhances liver fat oxidation, reduces liver fat synthesis, and increases adiponectin levels in animal models in vivo.

Recent reports suggest that NAFLD is associated with an increased risk of cardiovascular disease independent of associated cardiovascular risk factors. Furthermore type 2 diabetics and subjects with impaired glucose tolerance are characterized by an increase in both hepatic and myocardial fat and left ventricular (LV) dysfunction, particularly diastolic dysfunction. Myocardial steatosis is an independent predictor of diastolic dysfunction in type 2 diabetes mellitus as well as impaired glucose tolerance. However, the effect of saxagliptin therapy on liver and myocardial fat content, as well as LV systolic and diastolic function in patients with impaired glucose tolerance (IGT) or type 2 diabetes has not been previously studied. Recently, it has been demonstrated that myocardial triglyceride content is increased in type 2 diabetic patients and is associated with impaired left ventricular diastolic function, independently of age, body mass index (BMI), heart rate, visceral fat, and diastolic blood pressure. More recently, it has been shown that that obese normal glucose tolerant subjects, obese subjects with IGT, and type 2 diabetic subjects have increased myocardial fat compared to lean subjects. Thus, both IGT and type 2 diabetic subjects have increased myocardial steatosis and defects in LV function. GLP-1 has been shown to improve myocardial function and cardiac output in conscious chronically instrumented canine models of cardiac injury or heart failure. GLP-1 increased cardiac output and reduced left ventricular end diastolic pressure in association with reduced systemic vascular resistance, and it improved myocardial insulin sensitivity and myocardial glucose uptake in dogs with rapid pacing-induced dilated cardiomyopathy. However, no previous study has examined the effect of saxagliptin on myocardial fat or LV function in IGT or type 2 diabetic patients. Finally, the effect of saxagliptin on vascular inflammation and monocyte Nuclear Factor-KappaB (NFkappaB) remains to be studied. Patients with Impaired Glucose Tolerance (IGT)/ Impaired Fasting Glucose (IFG) have insulin resistance as a well established defect. Furthermore, as stated previously, both myocardial and hepatic steatosis as well as defects in LV function are well characterized in obese, insulin resistant patients with IGT. However, the effect of DPP IV inhibitors on hepatic and myocardial steatosis and monocyte inflammation in insulin resistant patients with IGT have not been previously studied.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a diagnosis diagnosis of Impaired Glucose Tolerance i.e. fasting plasma glucose less than or equal to 125 mg/dl, 2 hour post 75 gram oral glucose tolerance test (OGTT) plasma glucose between 140-199 mg/dl, glycosylated hemoglobin A1c (HbA1c) less than 6.5% as per American Diabetes Association (ADA) criteria.
* Women of childbearing potential (WOCBP) and men must be using an acceptable method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* Patients must not be on anti-diabetes therapy for treatment of Impaired Glucose Tolerance (IGT) and must have a fasting plasma glucose concentration less or equal to 125 mg/dl.
* Type 1 or Type 2 diabetes mellitus (fasting plasma glucose greater than 125 mg/dl).
* Patients must not be on or have received metformin, thiazolidinediones, sulfonylureas, DPP IV inhibitor, or exenatide/liraglutide treatment for treatment of IGT at any time. Patients must not be receiving any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications such as hormone replacement therapy with known adverse effects on glucose tolerance levels. Patients taking systemic glucocorticoids will also be excluded.
* Subjects with a history of clinically significant heart disease, peripheral vascular disease, or pulmonary disease.
* Subjects must have a Body Mass Index between 30-35 kg/m2 and stable body weight.
* Subjects must not have clinically significant liver disease (aspartate aminotransferase (AST) < 2.5 times upper limit of normal, Alanine transaminase (ALT) < 2.5 times upper limit of normal, Alkaline phosphatase< 2.5 times upper limit of normal), kidney disease (Serum creatinine < 1.5 mg/dl in men and 1.4 mg/dl in women) or significant anemia (Hematocrit < 34 vol%).
* Subjects with a history of any serious hypersensitivity reaction to saxagliptin or a dipeptidyl peptidase 4 (DPP-IV) inhibitor.
* Concomitant treatment with systemic cytochrome P450 3A4 inducers.
* Women who are pregnant or breastfeeding

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-02; Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Bajaj, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Saxagliptin: Saxagliptin 5 mg orally daily for 6 months
  Saxagliptin: Subjects will be randomized to receive either Saxagliptin 5mg daily orally or placebo for 6 months. All subjects will receive baseline measurements of fasting plasma glucose, free fatty acids, plasma adipocytokines, and plasma levels of inflammatory markers, plasma lipids, and glucose tolerance (75 gram oral glucose tolerance test) as well as measurement of liver and myocardial fat content and left ventricular systolic and diastolic function with magnetic resonance imaging/spectroscopy. All subjects will also undergo measurements of monocyte inflammatory proteins at baseline. All subjects will undergo repeat measurements of fasting plasma glucose, Free Fatty Acids, inflammatory markers and adipocytokines, oral glucose tolerance test, monocyte inflammation, as well as hepatic/myocardial fat content determination and left ventricular function at the end of the 6 months.
Period: Overall Study
Arm/Group | Placebo | Saxagliptin
Started | 4 | 4
Completed | 3 | 4
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Saxagliptin | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Myocardial and Hepatic Fat Content (Percentage)
Description: The percentage change in hepatic fat (%) and myocardial fat (%) from baseline as measured by magnetic resonance imaging and spectroscopy (MRS).
Time Frame: 6 months
Population: This data was not collected.
Groups:
- Saxagliptin: Saxagliptin 5 mg orally daily for 6 months
  Saxagliptin: Subjects will be randomized to receive either Saxagliptin 5mg daily orally or placebo for 6 months. All subjects will receive baseline measurements of fasting plasma glucose, free fatty acids, plasma adipocytokines, plasma levels of inflammatory markers and C Reactive Protein (CRP), Intracellular Adhesion Molecule (ICAM), vascular cell adhesion molecule (VCAM), plasma lipids, and glucose tolerance (75 gram oral glucose tolerance test) as well as measurement of liver and myocardial fat content and left ventricular systolic and diastolic function with magnetic resonance imaging/spectroscopy. All subjects will also undergo measurements of monocyte inflammatory proteins at baseline. All subjects will undergo repeat measurements of fasting plasma glucose, Free Fatty Acids, inflammatory markers and adipocytokines, oral glucose tolerance test, monocyte inflammation, as well as hepatic/myocardial fat content determination and left
Arm/Group | Placebo | Saxagliptin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)(%).
Description: The change in Left ventricular function measured as the percentage change in left ventricular ejection fraction (LVEF)(%) from baseline as measured by by magnetic resonance imaging.
Time Frame: 6 months
Population: This data was not collected.
Arm/Group | Placebo | Saxagliptin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Monocyte Inflammatory Protein NFkappaB(%)
Description: The percentage change in monocyte inflammatory proteins NFkappaB (%) from baseline.
Time Frame: 6 months
Population: This data was not collected.
Arm/Group | Placebo | Saxagliptin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Saxagliptin: Saxagliptin 5 mg orally daily for 6 months
  Saxagliptin: Subjects will be randomized to receive either Saxagliptin 5mg daily orally or placebo for 6 months. All subjects will receive baseline measurements of fasting plasma glucose, free fatty acids, plasma adipocytokines, plasma levels of inflammatory markersplasma lipids, and glucose tolerance (75 gram oral glucose tolerance test) as well as measurement of liver and myocardial fat content and left ventricular systolic and diastolic function with magnetic resonance imaging/spectroscopy. All subjects will also undergo measurements of monocyte inflammatory proteins at baseline. All subjects will undergo repeat measurements of fasting plasma glucose, Free Fatty Acids, inflammatory markers and adipocytokines, oral glucose tolerance test, monocyte inflammation, as well as hepatic/myocardial fat content determination and left
Arm/Group | Placebo | Saxagliptin
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT01548651/Prot_SAP_000.pdf